CLINICAL TRIAL: NCT05556434
Title: Machine Learning Algorithms Based on Clinical Data to Predict Postoperative Complications of Patients With Hepatolithiasis Undergoing Hepatectomy
Brief Title: Predicting Complications of Hepatolithiasis After Hepatectomy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Eastern Hepatobiliary Surgery Hospital (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Gang Chen, MD, Clinical Professor, Principal Investigator, First Affiliated Hospital of Wenzhou Medical University
Other Study IDs: prognosis of hepatolithiasis
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Liver Diseases; Complication
Keywords: liver resection; complication; risk factor; machine learning; hepatolithiasis
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with postoperative complications: Patients who experienced postoperative complications were divided into the first group. The complications were defined according to the Clavien-Dindo classification system.
  Interventions: Diagnostic Test: radiological evaluation
- patients without postoperative complications: Patients who didn't experience postoperative complications were divided into the second group.
  Interventions: Diagnostic Test: radiological evaluation

INTERVENTIONS:
Diagnostic Test: radiological evaluation — All patients undergoing hepatectomy receive imaging evaluation and laboratory test before and after surgery to define clinical parameters.
  diseases

SUMMARY:
Postoperative complications seriously affect the recovery of patients undergoing hepatectomy. Identifying risk factors and develop predictive models of complications for patients with hepatolithiasis undergoing hepatectomy is important for clinical practice.

DETAILED DESCRIPTION:
Along with the change of lifestyle and dietary habits, many people are diagnosed with hepatolithiasis that is especially prevalent in Asia. Liver resection remains the favorable curative therapy for hepatolithiasis with a relatively low recurrence rate. Although there have been great improvements in surgical techniques and perioperative management, postoperative complications remain commonplace and seriously threat the recovery of patients undergoing hepatectomy. Therefore, it is important to identify risk factors of complications to improve the overall prognosis of patients. We want to collect the clinical information of patients with hepatolithiasis undergoing hepatectomy, including demographic data , laboratory index, histological features and postoperative complications. Patients are followed up at a interval of 3 month after treatment, and the survival data and recurrence rate are recorded. Then the relationship between clinical data and short-term outcomes after surgery are explored. Then models based on clinical features are developed to predict short-term outcomes after hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* pathologically diagnosed hepatolithiasis
* without malignancies
* receiving liver resection
* Eastern Cooperative Oncology Group performance status (ECOG-PS) 0-2
* Child-Pugh score of ≤7
* complete clinical and follow-up information
* age between 18-80 years old

Exclusion Criteria:

* with malignancies
* receiving other treatments
* Eastern Cooperative Oncology Group performance status (ECOG-PS) >2
* Child-Pugh score of >7
* incomplete clinical data
* lost to follow up
* age <18 years old or >80 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatolithiasis who received liver resection for curative intent
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Complications | 3 months
  Postoperative complications and mortality are recorded according to the Clavien-Dindo classification system

SECONDARY OUTCOMES:
Recurrence of hepatolithiasis | 1 year
  Patients were followed-up at an interval of 3 months and recurrence of hepatolithiasis is evaluated by radiological methods.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Chen, MD,PhD, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- Gang Chen, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang T, Lau WY, Lai EC, Yang LQ, Zhang J, Yang GS, Lu JH, Wu MC. Hepatectomy for bilateral primary hepatolithiasis: a cohort study. Ann Surg. 2010 Jan;251(1):84-90. doi: 10.1097/SLA.0b013e3181b2f374. PMID 20032719
- [Background] Su CH, Shyr YM, Lui WY, P'Eng FK. Hepatolithiasis associated with cholangiocarcinoma. Br J Surg. 1997 Jul;84(7):969-73. doi: 10.1002/bjs.1800840717. PMID 9240138
- [Background] Tabrizian P, Jibara G, Shrager B, Schwartz ME, Roayaie S. Hepatic resection for primary hepatolithiasis: a single-center Western experience. J Am Coll Surg. 2012 Nov;215(5):622-6. doi: 10.1016/j.jamcollsurg.2012.07.005. Epub 2012 Aug 24. PMID 22921329
- [Background] Citterio D, Facciorusso A, Sposito C, Rota R, Bhoori S, Mazzaferro V. Hierarchic Interaction of Factors Associated With Liver Decompensation After Resection for Hepatocellular Carcinoma. JAMA Surg. 2016 Sep 1;151(9):846-53. doi: 10.1001/jamasurg.2016.1121. PMID 27248425
- [Background] Jarnagin WR, Gonen M, Fong Y, DeMatteo RP, Ben-Porat L, Little S, Corvera C, Weber S, Blumgart LH. Improvement in perioperative outcome after hepatic resection: analysis of 1,803 consecutive cases over the past decade. Ann Surg. 2002 Oct;236(4):397-406; discussion 406-7. doi: 10.1097/01.SLA.0000029003.66466.B3. PMID 12368667